CLINICAL TRIAL: NCT01860365
Title: Measuring Concerns and Needs of Cancer Patients Referred to Complementary Medicine Treatment Integrated Within the Oncology Service
Brief Title: Measuring Concerns of Cancer Patients Referred to Complementary Medicine Treatment Integrated Within Oncology Service
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Integrative oncology Program, Director, Carmel Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMC-09-0024-CTIL
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Quality of Life
Keywords: Quality of life; Integrative medicine; Supportive care; Cancer; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complementary medicine counseling (Experimental): Patients receiving chemotherapy who are referred by their oncology provider to complementary medicine consultation and treatment provided in addition to conventional supportive care
  Interventions: Other: Complementary medicine consultation and treatment
- Conventional supportive care (Active Comparator): Patients receiving conventional supportive care
  Interventions: Other: Patients receiving conventional supportive care

INTERVENTIONS:
Other: Complementary medicine consultation and treatment — Patients receiving chemotherapy will be referred by their oncology provider to complementary medicine (CM) consultation and treatment provided in addition to conventional supportive care.CM consultation will include assessment of patients' concerns and well-being, current CM use (including herbal and nutritional supplements), and construction of CM treatment based on efficacy and safety considerations.
  Arms: Complementary medicine counseling
Other: Patients receiving conventional supportive care — Patients receiving chemotherapy will be offered assessment of their concerns and well-being as well as their current complementary medicine (CM) use (including herbal and nutritional supplements). Patients in this arm study will receive conventional supportive care with no added CM consultation or treatment.
  Arms: Conventional supportive care

SUMMARY:
In 2007, the Haifa and Western Galilee district of the CHS set out to test the feasibility of integrating complementary medicine (CM) within the CHS Oncology Service. In 2008, the CHS established the Integrative Oncology Program with the goal of addressing patient concerns and improving quality of life parameters during chemotherapy and advanced disease. The study hypothesis is that integrated medicine consultation and treatment provided within the oncology department may improve patients' concerns and well-being.

DETAILED DESCRIPTION:
In 2007, the Haifa and Western Galilee district of the CHS set out to test the feasibility of integrating complementary medicine (CM) within the CHS Oncology Service. In 2008, the CHS established the Integrative Oncology Program with the goal of addressing patient concerns and improving quality of life parameters during chemotherapy and advanced disease. The study is purposed to assess concerns, needs and perspectives of patients referred to integrative consultation during chemotherapy and/or advanced cancer; to characterize social demographic and health parameters of patients who consult or avoid integrative medicine consultation; to document complementary medicine use prior and during consultation; to assess if complementary medicine consultation and treatment improve patient's concerns and well-being; and to assess oncology provider and integrative practitioner communications issues concerning integrative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer diagnosis receiving chemotherapy and/or surgical treatment who are referred by their oncology provider to complementary medicine consultation
* Age older than 18 years

Exclusion Criteria:

* Age younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2009-07; Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
MYCAW (Measure Yourself Concerns and Wellbeing)questionnaire | 6-12 weeks(+follow-up 4 months)
  Assessing patients'concerns and Wellbeing as well as narrative assessment of integrative care outcomes
ESAS (Edmonton Symptom Assessment Scale)questionnaire | 6-12 weeks(+follow-up 4 months)
  Assessing the severity of 10 leading symptoms and well-being
EORTC QLQ-C30 | 6-12 weeks(+follow-up 4 months)
  The EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the health related quality of life of cancer patients. The questionnaire includes functional and symptom scales.

SECONDARY OUTCOMES:
FACIT-Sp-12 questionnaire | 2-4 months
  Assessing patients' spiritual well-being
Attitudes concerning complementary medicine | 6-12 weeks
  Assessment of patients' attitudes concerning complementary medicine (CM)safety and efficacy, health beliefs concerning mind-body interactions, and willingness to receive CM treatments

OTHER OUTCOMES:
Complementary medicine side-effects documentation | 6-12 weeks(+follow-up 4 months)
  Documentation in registry protocol of patients' reported side-effects concerning complementary medicine treatments

CONTACTS AND LOCATIONS:
Overall Officials: Eran Ben-Arye, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Lin Zebulon and Carmel Medical centers, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hauzer M, Grimberg R, Samuels N, Keshet Y, Mordechai A, Dagash J, Ben-Arye E. Exploring primary care physician feedback following an integrative oncology consultation. Support Care Cancer. 2023 Oct 3;31(10):606. doi: 10.1007/s00520-023-08079-6. PMID 37787815
- [Derived] Ben-Arye E, Elly M, Gressel O, Reshef A, Shani Md M, Stein N, Saliba W, Samuels N. Exploring the effectiveness of a patient-tailored integrative oncology program on emotional distress during chemotherapy for localized cancer. Psychooncology. 2022 Feb;31(2):207-218. doi: 10.1002/pon.5794. Epub 2021 Aug 26. PMID 34435403
- [Derived] Kerner H, Samuels N, Ben Moshe S, Sharabi IS, Ben-Arye E. Impact of a patient-tailored complementary/integrative medicine programme on disturbed sleep quality among patients undergoing chemotherapy. BMJ Support Palliat Care. 2020 Sep;10(3):e21. doi: 10.1136/bmjspcare-2017-001351. Epub 2017 Jul 14. PMID 28710110
- [Derived] Sharabi IS, Levin A, Schiff E, Samuels N, Agour O, Tapiro Y, Lev E, Keinan-Boker L, Ben-Arye E. Quality of life-related outcomes from a patient-tailored integrative medicine program: experience of Russian-speaking patients with cancer in Israel. Support Care Cancer. 2016 Oct;24(10):4345-55. doi: 10.1007/s00520-016-3274-3. Epub 2016 May 11. PMID 27169571
- [Derived] Ben-Arye E, Keshet Y, Shahbar IM, Aharonson ML, Preis L, Agour O, Schiff E, Samuels N. The kitchen as therapy: qualitative assessment of an integrative cuisine workshop for patients undergoing chemotherapy. Support Care Cancer. 2016 Apr;24(4):1487-95. doi: 10.1007/s00520-015-2934-z. Epub 2015 Sep 11. PMID 26361759
- [Derived] Ben-Arye E, Samuels N, Schiff E, Raz OG, Sharabi IS, Lavie O. Quality-of-life outcomes in patients with gynecologic cancer referred to integrative oncology treatment during chemotherapy. Support Care Cancer. 2015 Dec;23(12):3411-9. doi: 10.1007/s00520-015-2690-0. Epub 2015 Mar 10. PMID 25752885